CLINICAL TRIAL: NCT01619878
Title: An Open-label, Single-arm Study to Evaluate the Efficacy, Safety and PK of Artemether-lumefantrine Dispersible Tablet in the Treatment of Acute Uncomplicated Plasmodium Falciparum Malaria in Infants <5 kg Body Weight
Brief Title: Efficacy, Safety and Pharmacokinetics of Artemether-lumefantrine Dispersible Tablet in the Treatment of Malaria in Infants < 5 kg
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCOA566B2306; 2011-005852-33; 2011-005858-33 (Other: Eudra CT)
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Results first posted 2015-06-17 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Acute Uncomplicated Falciparum Malaria
Keywords: plasmodium; P. falciparum; malaria; infant; neonate
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

ARMS (1):
- Cohort 1 (Experimental): One Artemether-lumefantrine (COA566) dispersible tablet taken orally twice a day during 3 days.
  Infants age >28 days.
  Interventions: Drug: Artemether-lumefantrine (COA566)

INTERVENTIONS:
Drug: Artemether-lumefantrine (COA566) — One dispersible tablet taken orally twice a day during 3 days.
  Other Names: Artemether-lumefantrine, COA566

SUMMARY:
The purpose of the study is to obtain efficacy, safety and pharmacokinetic (PK) data following treatment with artemether-lumefantrine dispersible tablet in infants < 5 kg of body weight (BW) with uncomplicated falciparum malaria.

ELIGIBILITY:
Inclusion Criteria:

* Neonates / infants
* Body weight < 5 kg
* In cohort 1, infants aged > 28 days; in cohort 2, neonates of a term age 0 to ≤ 28 days
* Microscopically confirmed diagnosis of acute uncomplicated Plasmodium falciparum malaria or mixed infections with an asexual Plasmodium falciparum parasitaemia of > 1,000 and < 100,000 parasites/µL

Exclusion Criteria:

* Presence of severe malaria (according to World Health Organization definition)
* Presence of the following signs of a critical condition: apnea-bradycardia, sustained bradycardia, tachycardia, desaturation, hypotension, hypothermia; or other severely deteriorated general condition (based on IMCI criteria in sick infants)
* Presence of any clinically significant neurological condition
* Presence of clinically significant abnormality of the hepatic and renal systems
* Patients who sustained a significant blood volume loss (> 3% of calculated blood volume) in the past 30 days
* Patients unable to swallow or whose drinking is impaired
* Family history of congenital prolongation of the QTc interval or sudden death or with any other clinical condition known to be associated with prolongation of the QTc interval such as history of symptomatic cardiac arrhythmias, with clinically relevant bradycardia or with severe cardiac disease
* Disturbances of electrolyte balance (e.g. hypokalaemia or hypomagnesaemia)
* Presence of any age-adjusted clinically or hematologically relevant laboratory and blood chemistry abnormalities
* Other protocol-defined inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Benin (2):
  - Novartis Investigative Site, Cotonou
  - Novartis investigative site, Cotonou
- Burkina Faso (2):
  - Novartis Investigative Site, Burkina Faso
  - Novartis investigative site, Ouagadougou
- Novartis investigative site, Calabar, Nigeria
- Novartis investigative site, Kinshasa, Republic of the Congo
- Novartis investigative site, Lomé, Togo

REFERENCES:
- [Derived] Tiono AB, Tinto H, Alao MJ, Meremikwu M, Tshefu A, Ogutu B, Ouedraogo A, Lingani M, Cousin M, Lefevre G, Jain JP, Duparc S, Hamed K. Increased systemic exposures of artemether and dihydroartemisinin in infants under 5 kg with uncomplicated Plasmodium falciparum malaria treated with artemether-lumefantrine (Coartem(R)). Malar J. 2015 Apr 15;14:157. doi: 10.1186/s12936-015-0682-7. PMID 25886021

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participant that did not complete in the "6 week follow-up phase" was also included in "Follow-up at 12 Months of Age" and was lost to follow-up
Period: 6 Week Follow-up Phase
Arm/Group | Cohort 1
Started | 20
Completed | 19
Not Completed | 1
Not completed — Adverse Event | 1
Period: Follow-up at 12 Months of Age
Arm/Group | Cohort 1
Started | 20
Completed | 17
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cohort 1
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: days] | 99.1 (51.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Polymerase Chain Reaction (PCR) Corrected 28 Day Parasitological Cure Rate
Description: Number of participants with clearance of asexual parasites by day 7 after initiating study treatment without recrudescence at day 28, corrected for re-infection by Polymerase Chain Reaction (PCR) assay.
Time Frame: 28 days
Population: Full analysis set (FAS) - all subjects receiving at least one dose of study drug and who are confirmed to have P. falciparum malaria at baseline.
Measure: Number; unit: number of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 20
number of participants | 16

2. Secondary Outcome: Polymerase Chain Reaction (PCR) Corrected Parasitological Cure Rate at Day 14 and 42
Description: Number of participants with clearance of asexual parasites by day 7 after initiating study treatment without recrudescence at day 14 and day 42, corrected for re-infection by Polymerase Chain Reaction (PCR) assay.
Time Frame: Day 14 and 42
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 20
Number of participants
  Day 14 | 16
  Day 42 | 16

3. Secondary Outcome: Number of Participants With Parasitological Uncorrected Cure Rate at Day 3, 7, 14, 28 and 42
Description: Number of patients with clearance of asexual parasites at day 3, 7, 14, 28 and 42 after initiating study treatment.
Time Frame: Day 3, 7, 14, 28 and 42
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 20
participants
  Day 3 | 20
  Day 7 | 16
  Day 14 | 16
  Day 28 | 10
  Day 42 | 7

4. Secondary Outcome: Percent Change of Parasite Count From Baseline at 24 Hours
Description: Percent change of parasite count from baseline at 24 hours
Time Frame: baseline, 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Cohort 1
Number analyzed (Participants) | 20
Percent Change | -99.4 (1.19)

5. Secondary Outcome: Number of Participants With Parasitaemia at 48 Hours After Treatment Initiation Greater Than at Baseline
Description: Number of participants with parasite density at 48 hours after treatment initiation greater than parasite density at baseline.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 20
participants | 0

6. Secondary Outcome: Number of Participants With Parasitaemia at 72 Hours After Treatment Initiation Greater Than or Equal to 25 Percent of Count at Baseline
Description: Number of participants with parasite density at 72 hours after treatment initiation greater than or equal to 25 percent of parasite density at baseline.
Time Frame: 72 hours
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 20
participants | 0

7. Secondary Outcome: Time to Parasite Clearance (PCT)
Description: Time from first dose until first total and continued disappearance of asexual parasite forms which remains at least a further 48 hours.
Time Frame: Up to 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1
Number analyzed (Participants) | 20
hours | 29.1 (9.6)

8. Secondary Outcome: Time to Fever Clearance (FCT)
Description: Time from first dose to the first time the axillary body temperature decreased below and remained below 37.5° C for at least 48 hours.
Time Frame: Up to 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1
Number analyzed (Participants) | 20
hours | 4.02 (6.433)

9. Secondary Outcome: Time to Gametocyte Clearance (GCT)
Description: Time from first dose until first total and continued disappearance of gametocytes which remains at least a further 48 hours.
Time Frame: Up to 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1
Number analyzed (Participants) | 20
hours | 36.32 (77.294)

ADVERSE EVENTS:
Arm/Group | Cohort 1
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=20)
Anaemia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Cerebral malaria (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=20)
Anaemia (Blood and lymphatic system disorders) | 6
Enteritis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Pyrexia (General disorders) | 5
Bronchitis (Infections and infestations) | 6
Gastroenteritis (Infections and infestations) | 2
Malaria (Infections and infestations) | 11
Rash pustular (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.